CLINICAL TRIAL: NCT03227276
Title: Double-blind, Randomised, Placebo-controlled 1-year Study to Evaluate the Efficacy and Safety of Litramine in Reducing Body Weight in Overweight and Moderately Obese Subjects
Brief Title: Efficacy and Safety of Litramine in 1 Year Weight Loss Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/004317
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Excess Calories; Overweight and Obesity; Weight Loss
Keywords: Litramine; Opuntia ficus-indica; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo tablet
- Litramine (Experimental)
  Interventions: Dietary Supplement: Litramine

INTERVENTIONS:
Dietary Supplement: Litramine — 2 tablets to be taken 3 times a day after meals
  Arms: Litramine
Dietary Supplement: Placebo tablet — 2 tablets to be taken 3 times a day after meals
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Litramine in reducing body weight in the context of an energy-restricted diet in overweight and moderately obese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 70 years old
2. Overweight (BMI 25 kg/m2 - 29.9 kg/m2) for 80% of randomized subjects and obese (BMI 30 kg/m2 - 34.9 kg/m2) for 20% of randomized subjects
3. Generally in good health
4. Desire to lose weight
5. Readiness and ability to complete the 1-year study, according to investigator's judgement following the screening interview
6. Accustomed to regular daily consumption of 3 main meals (breakfast, lunch, dinner)
7. Consistent and stable body weight in the last 3 months prior to V1 (less than 5% self- reported change)
8. Subject's agreement to comply with study procedures, in particular:

   * to take IP as recommended
   * to avoid the use of other weight loss and/or management products and/or programs during the study
   * to adhere to diet recommendation during the study
   * to complete the subject diary and study questionnaires
9. Women of childbearing potential:

   * commitment to use contraception methods
   * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
10. Written informed consent

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational products or source plants
2. Pathological electrocardiogram (ECG) at V1
3. History and/or presence of clinically significant condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   * untreated or unstable thyroid gland disorder
   * untreated or unstable hypertension (regular blood pressure >140/90 mm Hg)
   * acute or chronic gastrointestinal (GI) disease or digestion/absorption disorders (e.g.

   inflammatory bowel disease, coeliac disease, pancreatitis etc.)
   * diabetes mellitus type 1
   * untreated or unstable diabetes mellitus type 2
   * any other serious organ or systemic diseases that could influence the conduct and/or outcome of the study and/or could affect the tolerability of the subject
4. Significant surgery within the last 6 months prior to V1:

   * GI surgery
   * liposuction
5. History of eating disorders like bulimia, anorexia nervosa, binge-eating within the last 12 months prior to V1
6. Deviation of safety laboratory parameter(s) at V1 that is:

   * clinically significant or
   * >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
7. Any electronic medical implant
8. Regular medication and/or supplementation and/or treatment within the last 3 months prior to V1 and during the study:

   * that could influence body weight (e.g. systemic corticosteroids)
   * that could influence gastrointestinal functions (e.g. laxatives, opioids, anticholinergics etc.) as per investigator judgement
   * for weight management (e.g. fat binder, carbohydrate/starch blocker, fat burner, satiety products, acupuncture etc.)
9. Smoking cessation within 6 months prior to V1 or during the study (regular smoking during the study at the same level as prior to the study is allowed)
10. Women of child-bearing potential: pregnancy or nursing
11. History of or current abuse of drugs, alcohol or medication
12. Participation in another clinical study in the 30 days prior to V1 and during the study
13. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Difference in mean body weight (kg) of overweight subjects | 52 weeks
  Difference in mean body weight (kg) of overweight subjects after 52 weeks of IP intake in comparison between verum and placebo

SECONDARY OUTCOMES:
Difference in mean body weight (kg) of all subjects | 52 weeks
Difference in mean body weight (kg) of obese subjects | 52 weeks
Proportion of subjects who lost at least 3%, 5% and 10% of baseline body weight | 52 weeks

OTHER OUTCOMES:
Adverse effects | 52 weeks
  Assessment of adverse events throughout the study
Safety parameters (Lab parameters, vital signs) | 52 weeks
  Assessment of laboratory results in full blood count, clinical chemistry, blood pressure and pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bongartz, MD, Principal Investigator — Analyze & Realize
Locations (1):
- Analyze & Realize, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided